CLINICAL TRIAL: NCT05595772
Title: PRGF VS CGF in Management of Labial Dehiscence Around Immediate Implants (Comparative Study) {PRGF= Plasma Rich in Growth Factors } {CGF=Concentrated Growth Factor}
Brief Title: Comparison of Two Different Types of Platelet Concentrate to Augment Bone Around Immediate Dental Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hussein Fathy Mohammad Hussein Abo Elkheir, Principal Investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HFMHAElkhe0001
Record Dates: First submitted 2022-10-13; First posted 2022-10-27 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Dental Implant Failure Nos
Keywords: immediate implant; PRGF; CGF; Plasma rich in growth factors; concentrated growth factor; labial dehiscence; platelet concentrate; bio-membrane; xenogenic bone graft
MeSH Terms: interventions — Intercellular Signaling Peptides and Proteins; Tooth Extraction

STUDY DESIGN:
Intervention Model Description: The study will use simple randomization to allocate patients into 2 groups, each group will be included 10 patients.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Concentrated Growth Factor) CGF (Active Comparator): ten patients indicated for immediate implant in the maxillary anterior region (class II socket)
  Interventions: Drug: Drug: Growth Factors (CGF); Procedure: Surgery: Dental Implant surgery; Procedure: Tooth extraction; Procedure: Xenogenic bone grafting
- group B (Plasma Rich in Growth Factor) PRGF (Active Comparator): Ten patients who indicated immediate implant in the maxillary anterior region (class I or class II socket),
  Interventions: Drug: Drug: Growth Factors (PRGF); Procedure: Surgery: Dental Implant surgery; Procedure: Tooth extraction

INTERVENTIONS:
Drug: Drug: Growth Factors (CGF) — Application of biological membrane of Concentrated growth factor (CGF) over bone grafting and implant
  Other Names: Concentrated growth factor
  Arms: group A (Concentrated Growth Factor) CGF
Drug: Drug: Growth Factors (PRGF) — Application of biological membrane of Plasma rich in growth factors combined with Xenogeneic bone grafting material around immediate implant
  Other Names: Plasma rich in growth factors
  Arms: group B (Plasma Rich in Growth Factor) PRGF
Procedure: Surgery: Dental Implant surgery — Immediate implant following extraction
Procedure: Tooth extraction — A Traumatic tooth extraction
Procedure: Xenogenic bone grafting — Application of bovine bone grafting over area of dehiscence around immediate implant
  Arms: group A (Concentrated Growth Factor) CGF

SUMMARY:
The goal of this clinial trial is to detect Which one of two different platelet concentrate bio-membrane (first or third generation) is better in terms of marginal bone level and bone density around immediate implants in esthetic zone using Cone beam computerized tomography The plasma rich in growth factor or concentrated growth factor?

20 patients with nonrestorable maxillary tooth in the esthetic zone, Subjects will be enrolled

The study will use simple randomization to allocate patients into 2 groups, each group will be included 10 patients: Group A: (concentrated growth factor group) ten patients indicated for immediate implant in the maxillary anterior region (class II socket), will be a candidate for immediate implant placement with CGF combined with xenogeneic bone graft Group B: (platelet-rich in growth factor group) Ten patients who indicated immediate implant in the maxillary anterior region (class I or class II socket), will be a candidate for immediate implant placement with PRGF combined with xenogeneic bone graft.

DETAILED DESCRIPTION:
with the increasing practice of dental implants; the esthetic outcome is considered as important as the functional and biological outcome Immediate implants have been evolved as the first treatment option in cases of the failed tooth to decrease the time of treatment plan To obtain an effective esthetic outcome with a single implant-supported restoration in the anterior region, it is crucial to preserve and maintain intact the bone anatomy

Numerous studies have explored the suitability of biocompatible materials in regenerative medicine. Platelet concentrates are originated from centrifuged blood and are named according to their biological characteristics, such as platelet-rich plasma, platelet-rich fibrin, and concentrated growth factor

Plasma rich in growth factors (PRGF), a subtype of P-PRP (pure platelet-rich plasma), is a supernatant enriched in plasma and platelet-derived morphogens, proteins, and growth factors. PRGF represents a complex pool of active mediators that may stimulate and accelerate tissue regeneration, which is generally safe to use and economical to obtain. Autologous PRGF has been approved for clinical use by the European Community and the U.S. Food and Drug Administration

CGF (concentrated growth factor), the third-generation platelet concentrate presented by Sacco in 2006 carries more growth factors and has a firmer fibrin structure than first-generation PRP and second-generation PRF (platelet-rich fibrin)

Aim of the study is

1. : Assess the effectiveness of PRGF and CGF in the management of buccal dehiscence and marginal bone level around the immediate implant.
2. : Compare the effectiveness of PRGF Vs CGF.

20 patients with nonrestorable maxillary tooth in the esthetic zone, Subjects will be enrolled

The study will use simple randomization to allocate patients into 2 groups, each group will be included 10 patients: Group A: (concentrated growth factor group) ten patients indicated for immediate implant in the maxillary anterior region (class II socket), will be a candidate for immediate implant placement with CGF combined with xenogeneic bone graft Group B: (platelet-rich in growth factor group) Ten patients who indicated immediate implant in the maxillary anterior region (class I or class II socket), will be a candidate for immediate implant placement with PRGF combined with xenogeneic bone graft.

Protocol for CGF preparation:

10 ml venous blood samples will be drawn from the patients and placed in a centrifuge tube without anticoagulants. Then the tubes will be placed in the centrifugation device in an opposing balanced manner and rotated in four sequential steps. The first step at 735 g (2249 ≈ 2200) for 2 min., the second one at 580 g (1998 ≈ 2000) for 4 min., the third one at 735 g (2249 ≈ 2200) for 4 min. and the fourth one at 905 g (2495 ≈ 2500) for 3 min. The result was a clot that was collected using a straight tweezer and ready to be used

Protocol for PRGF preparation:

30 ml venous blood will be collected from the patient then deposited in 5 mL tubes containing sodium citrate anticoagulant. Then the tubes will be centrifuged at 580 G (2270 rpm) for 8 minutes at room temperature. After centrifugation, the blood sample will be layered into the following four distinctive layers:

1. 0.5 mL Plasma poor in growth factors (PPGFs) =F1 in the uppermost part of the tube
2. 0.5 mL Plasma with growth factors (PGFs) = F2
3. 0.5 mL (PRGF) = F3 located immediately above the red blood cell portion in the tube
4. Red blood cell concentrate layer From all tubes, The 500 μL PPGF will be eliminated and the PRGF will be separated with 500 μL pipettes and transported to an independent dish then activated using 50 μL of 10% calcium chloride for every 1 ml of preparation and mixed with xenogenic bone graft then it will be incubated for 40 minutes in 37̊c to produce easy to handle gelatinous layer (PRGF) fibrin mixed with the xenogenic bone.

Surgical Phase

1. The surgical site will be prepared by scrubbing the surgical site using Betadine: Povidone-iodine, 7.5% (0.75% available iodine) the Nile Comp. for Pharmaceuticals and Chemical Industries, Alexandria, Egypt
2. Nerve block or infiltration anesthesia will be administrated Articaine (4%) with epinephrine (1:100,000 or 1:200,000)
3. Atraumatic extraction of the tooth or remaining root using periotome, then sequential implant drilling accompanied by copious irrigation will be carried out. then cover screw attached to the implant top by the aid of its driver
4. A sample of venous blood will be withdrawn from the patient and centrifuged without delay according to the preparation protocol of each group.
5. Then the membrane loaded with the bone graft will be applied and condensed around the dental implant filling the gap between the fixture and the walls of the socket.
6. Finally, Tension-free Closure of the wound was achieved using 4/0 vicryl sutures.

ELIGIBILITY:
Inclusion Criteria:

1. Selected patients of both sexes are 20-40 years old.
2. Patients are systemically healthy based on questionnaire dental modification of Cornell index.
3. Gingival health according to the new classification system (2017)
4. The recipient site of the implant is free from any pathological conditions.
5. Class II extraction socket according to Chang's classification system
6. Adequate interocclusal space to accommodate the available restorative components.
7. Adequate native/apical bone to achieve primary implant stability.

Exclusion Criteria:

1. Pregnant female.
2. Para-functional habits such as bruxism and clenching Patients suffering from periodontitis.
3. Smokers.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Bone density | 9 months
  evaluation of bone density around immediate implants as (D1,D2,D3,D4)
Marginal bone level. | 9 months
  evaluation of marginal bone level around implant in comparison with baseline bone level immediately after surgery using a fixed point on CBCT

CONTACTS AND LOCATIONS:
Overall Officials: ahmed a khalil, PhD, Study Director — oral medicine and periodontology department faculty of dentistry minia university; Ahmed a Mustafa, PhD, Study Director — oral medicine and periodontology department faculty of dentistry minia university; hussein f mohammad, bachelor, Principal Investigator — oral medicine and periodontology department faculty of dentistry minia university
Locations (1):
- Faculty of Dentistry Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
age medical history oral hygiene status
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after study completion and for 3 years
Access Criteria: investigators related to official organization